CLINICAL TRIAL: NCT00214773
Title: MPS VI Clinical Surveillance Program (CSP)
Brief Title: Mucopolysaccharidosis (MPS) VI Clinical Surveillance Program (CSP)
Status: Completed | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: MPSVI CSP
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2019-01

CONDITIONS: Mucopolysaccharidosis VI (MPS VI, Maroteaux-Lamy Syndrome)
MeSH Terms: conditions — Mucopolysaccharidosis VI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: No intervention. This is an observational program.

SUMMARY:
The objectives of this program are: to further characterize the natural progression of MPS VI disease; to generate and disseminate information on the care and management of MPS VI patients to clinical and medical professionals; to provide a resource to physicians and patients by providing information for optimizing patient care based on aggregate data; to characterize the clinical response to long-term Naglazyme® (galsulfase) treatment; to further characterize the long-term safety of Naglazyme® treatment.

ELIGIBILITY:
Inclusion Criteria

All patients must meet the following criteria to qualify for enrollment in the CSP:

* Patient or patient's parent or legal guardian, if child is under 18 year old or is unable to consent, has provided a signed Patient Information and Authorization Form.
* Patient has laboratory results confirming a diagnosis of MPS VI disease based on detection of deficient ARSB activity (on fibroblasts, leucocytes or dried blood spots)and/or abnormality on the ARSB gene.
* Patient is willing to undergo general assessments to establish baseline data or permits physician to enter assessment data recorded prior to CSP entry if available in the patient's medical records. General assessments include: urinary GAG level, urinary protein level, serum sample for antibody levels, height, weight, and patient history.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a confirmed diagnosis of MPS VI disease may participate in the CSP. It is not a requirement that the patients enrolled in the CSP receive Galsulfase 1mg/kg to participate as this is an observational program.
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2005-07; Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
To further characterize the natural progression of MPS VI disease, irrespective of treatment modality and to evaluate efficacy and safety treatment with Galsulfase. | at least 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Julie Johnson, Study Director — BioMarin Pharmaceutical
Locations (50):
- United States (23):
  - University of California, Irvine, Irvine, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Emory University, Decatur, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Baton Rouge Clinic, Baton Rouge, Louisiana
  - Tulane University Medical Center, New Orleans, Louisiana
  - Johns Hopkins Univeristy School of Medicine, Baltimore, Maryland
  - Children's Health Care, Minneapolis, Minnesota
  - University of Minnesota - Fairview University Medical Center, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - St. Joseph's Healthcare, Paterson, New Jersey
  - New York University, New York, New York
  - Fullerton Genetic Center, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Sioux Valey Children's Speciality Clinics, Sioux Falls, South Dakota
  - University of Utah Medical Center, Salt Lake City, Utah
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Australia (5):
  - Westmead Hospital, Wentworthville, New South Wales
  - Royal Children's Hospital, Brisbane, Brisbane, Queensland
  - Women and Children's Hospital, Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Subiaco, Western Australia
- LKH-Universitätsklinik Graz, Kinderklinik, Graz, Styria, Austria
- Institute of Pathology and Genetics, Metabolic Unit, Charleroi, Wallonia, Belgium
- France (2):
  - Hôpital Femme Mère Enfant, Bron, Auvergne-Rhône-Alpes
  - Hopital Necker - Enfants Malades, Paris
- Germany (5):
  - Oberarzt Pädiatrie, Hanover, Lower Saxony
  - Universitatsklinikum Freiburg, Klinik II, Kammin, Mecklenburg-Vorpommern
  - Universitätsmedizin, Mainz, Rheinland-Pfalz RP
  - Charité-Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
- MidWestern Regional Hospital, Limerick, Ireland
- Italy (3):
  - Azienda Ospedaliero Universitaria, Cibali, Catania
  - Department of Woman's and Child's Health, Padua, Veneto
  - Università Milano Bicocca, Resp. Centro "Fondazione Mariani", Monza
- Vilnius University Hospital, Santariskiu Klinikos, Vilnius, Lithuania
- Rotterdam University Hospital - Sophia's Children's Hospital, Rotterdam, Netherlands
- Hospital de Sao Joao, Unidae de Doencas Metabolicas, Porto, Portugal
- Astrid Lindgrens Children's Hospital, Stockholm, Sweden
- United Kingdom (5):
  - Queen Elizabeth Hospital, University Hospitals Birmingham NHS, Birmingham
  - Birmingham Children's Hospital, Steelhouse, Birmingham
  - Great Ormond Street Hospital For Children, NHS Foundation Trust, London
  - St Mary's Hospital, Willink Biochemical Genetics Unit, Manchester
  - Salford Royal Hospital NHS Trust, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Solanki GA, Sun PP, Martin KW, Hendriksz CJ, Lampe C, Guffon N, Hung A, Sisic Z, Shediac R, Harmatz PR; CSP Study Group. Cervical cord compression in mucopolysaccharidosis VI (MPS VI): Findings from the MPS VI Clinical Surveillance Program (CSP). Mol Genet Metab. 2016 Aug;118(4):310-8. doi: 10.1016/j.ymgme.2016.06.001. Epub 2016 Jun 3. PMID 27339555
- See also: BioMarin Pharmaceutical Inc Website — http://www.BRMN.com